CLINICAL TRIAL: NCT02923388
Title: Neuroprotective Effect of Vitamin B12 and Vitamin B6 Against Vincristine Induced Peripheral Neuropathy: A Randomized, Double Blind, Placebo Controlled, Multi Center Trial
Brief Title: Neuroprotective Effect of Vitamin B12 and Vitamin B6 Against Vincristine Induced Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Fatiha Tasmin Jeenia, Resident, Department of Pharmacology, BSMMU, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: No. BSMMU/2016/8305
Record Dates: First submitted 2016-08-31; First posted 2016-10-04 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Vincristine Induced Peripheral Neuropathy (VIPN)
MeSH Terms: interventions — Vitamin B 12; Vitamin B 6; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Active Comparator): Intervention: Injection Mecobalamin (500mcg) three times a week (day 1, 3 and 5 of vincristine chemotherapy) for 5 weeks.
  Intervention: Tablet Pyridoxine hydrochloride (25 mg) 2 tablets thrice daily for 5 weeks.
  Interventions: Drug: Injection Mecobalamin,; Drug: Tablet Pyridoxine hydrochloride
- Placebo (Placebo Comparator): Intervention: Injection normal saline (1 ml) three times a week (day 1, 3 and 5 of vincristine chemotherapy) for 5 weeks.
  Intervention: Oral placebo pill 2 tablets thrice daily for 5 weeks.
  Interventions: Drug: Intravenous normal saline 1 ml; Drug: Placebo pill

INTERVENTIONS:
Drug: Injection Mecobalamin, — Injection Mecobalamin (500mcg) three times a week (day 1, 3 and 5 of vincristine chemotherapy) for 5 weeks.
  Other Names: Vitamin B12
  Arms: Experimental
Drug: Tablet Pyridoxine hydrochloride — Tab. Pyridoxine hydrochloride (25 mg) 2 tablets thrice daily for 5 weeks
  Other Names: Vitamin B6
  Arms: Experimental
Drug: Intravenous normal saline 1 ml — Normal saline 1 ml three times a week (day 1, 3 and 5 of vincristine chemotherapy) for 5 weeks
  Other Names: Normal saline
  Arms: Placebo
Drug: Placebo pill — Placebo pill orally thrice daily for 5 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This study will be conducted to evaluate the effect of vitamin B12 and vitamin B6 in delaying the onset and reducing the incidence and severity of Vincristine Induced Peripheral Neuropathy (VIPN) in Acute Lymphoblastic Leukemia (ALL) patient.

DETAILED DESCRIPTION:
Acute Lymphoblastic Leukemia (ALL) is an emerging health burden for Bangladesh. It is anticipated that about 20 million people are going to be affected annually by 2025 in countries currently on developmental transition. Good prognostic outcome of ALL relies on uninterrupted and complete course of chemotherapy. About 85% of adult patients and 98% of children attain complete recovery with full course of treatment. One of the crucial chemotherapeutic agents used to treat ALL is vincristine. It is needed to complete vincristine with adequate dose in order to get a better prognostic outcome. About 45% of the patients getting vincristine develop a deleterious side effect called Vincristine Induced Peripheral Neuropathy (VIPN). Unfortunately, development of VIPN results in dose reduction, protocol deviation and even abandonment of treatment with vincristine in some ALL patients. Better prognostic outcome becomes an arcadia. So far, many researches have been conducted to explore a way to prevent or treat VIPN. But still no conclusive recommendation can be made. Therefore, VIPN has become an important issue need to be addressed. This study will be a small effort to identify the potential of vitamin B12 and vitamin B6 as probable preventive measures of VIPN. Evidence suggests that, vitamin B12 and vitamin B6 two water soluble, non toxic vitamins well recognized for the treatment of peripheral neuropathy. Vitamin B12 plays a very fundamental role in neurological function. It exerts its physiological effects through mediating two principal enzymatic pathways by which it maintains the integrity of neuronal membrane. On the other hand, vitamin B6 or pyridoxine is an essential co- factor in various synthesis pathways including synthesis of myelin sheath. Patients will be randomly allocated into two arms by using online research randomizer and newly diagnosed ALL patients will be enrolled in this research. From the day of starting chemotherapy, patients on arm A (Intervention arm) will be concurrently administered with vitamin B12 and vitamin B6. Vitamin B12 will be given 500 μg three times a week intravenously on a basis of every alternate day except the day of receiving vincristine and vitamin B6 will be given 50 mg thrice daily orally during the induction period (5 weeks) of chemotherapy cycle. On the other hand, patients on arm B (Placebo arm) will be given placebo pill and intravenous placebo injection at same interval. Prior to initiation of induction chemotherapy each participant will undergo neuropathy evaluation per National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.0 scale and will be interviewed according to the neurotoxicity subscale of Functional Assessment of Cancer Therapy (FACT) -GOG- Ntx quality of life assessment questionnaire. The participants will be re-evaluated once weekly on the outset of 2nd week, 3rd week, 4th and 5th week of vincristine chemotherapy during induction period. They will be assessed per NCI-CTCAE v.4.0 scale for severity of neuropathy and by FACT- GOG- Ntx by answering specific questions regarding the presence of tingling, numbness, pain, muscle weakness and motor activities. As neuropathy and neuropathic pain are mostly subjective issue rather than objective and reflected more comprehensively by the particular person encountering with, so patient based measures will be used in this study. Incidence, onset and severity of peripheral neuropathy will be compared on both arms.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older with newly diagnosed ALL going to start induction chemotherapy with Vincristine
2. Patients with good performance status (ECOG 0- 3)
3. Patients with no preexisting peripheral neuropathy
4. Patients with grade 0 neuropathy on admission
5. Patients with normal renal function (Serum creatinine <1.5 mg/dl)
6. Patients agree to participate in the study signing an informed written consent

Exclusion Criteria:

1. Pregnant women and nursing mothers
2. Patients with clinical neuropathy due to diabetes mellitus or other causes
3. Patients with head neck tumors
4. Patients taking anticonvulsants, antidepressants, opioids, vitamin E and other neuropathic pain medication agents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Time of onset of Vincristine Induced Peripheral Neuropathy | 0 weeks (baseline), change in neuropathy status on the outset 2nd week, 3rd week, 4th week and 5th week of vincristine chemotherapy
Severity of Vincristine Induced Peripheral Neuropathy | On the outset of 1st week change in the severity of neuropathy on the outset of 2nd week, 3rd week, 4th week, 5th week of vincristine chemotherapy
Incidence of Vincristine Induced Peripheral Neuropathy | Cumulative incidence at 5th week of vincristine chemotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Bangabandhu Sheikh Mujib Medical University, Dhaka
  - Dhaka Medical College Hospital, Dhaka

IPD SHARING:
Plan to Share IPD: No